CLINICAL TRIAL: NCT02080325
Title: Vegetarian High Protein Weight Loss Diets
Acronym: ALPROsoya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 783 Soya; ALPRO™ Foundation (Other Grant/Funding Number: The Scottish Government's Rural and Environment Science and Analytical Services Division)
Record Dates: First submitted 2014-02-28; First posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Obesity
Keywords: weight loss; high protein diet; plant protein; satiety; soy
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Protein-Weight loss-Meat/High Protein-Weight loss Soy (Other): After 3 Days - Normal Protein Maintenance diet (NP- MTD, 3 days), there is the first arm of the study, Days 14 days- randomised to High Protein-Weight loss-Meat with High Protein-Weight loss-Soy
  Interventions: Other: High Protein-Weight loss-Soy diet; Other: High Protein-Weight loss-Meat
- High Protein-Weight loss-Soya/High Protein Weight loss-meat (Other): After 3 Days - Normal Protein Maintenance diet (NP- MTD, 3 days), there is the first arm of the study, Days 14 days- randomised to High Protein-Weight loss-Soy with High Protein-Weight loss-Meat
  Interventions: Other: High Protein-Weight loss-Soy diet; Other: High Protein-Weight loss-Meat

INTERVENTIONS:
Other: High Protein-Weight loss-Soy diet — • The high protein (HP) weight loss diet will be fed to 100% resting metabolic rate (RMR) on a 5 day rotation menu, fed as three meals a day, 30% protein, 30% fat and 40% carbohydrate; the soya version based on soya protein or soya-tvp (textured vegetable protein).
  Other Names: SOY HP WL diet
Other: High Protein-Weight loss-Meat — • The high protein (HP) weight loss diet will be fed to 100% resting metabolic rate (RMR) on a 5 day rotation menu, fed as three meals a day, 30% protein, 30% fat and 40% carbohydrate; the meat version will be based on chicken and beef meat.
  Other Names: MEAT HP WL diet

SUMMARY:
This study aims to investigate the mechanistic processes involved in protein-induced satiety/satiation during weight loss in humans.

Thsi study will investigate:

* How do high-protein weight loss (HPWL) diets rich in meat or soya based protein sources impact on profile of 'motivation to eat' both within a day and between days ?
* Do biomarkers of satiety alter differentially on meat or soya HPWL diet, as measured by monitoring alteration in plasma amino acids and gut-related hormones ?
* How does a vegetarian and meat-based weight loss diet impact on nitrosamine excretion in faecal samples, as an indicator of faecal toxicity?

Previous work has indicated that high-protein (30% protein) weight loss diets are more satiating (produce less hunger) than normal protein WL diet (15% protein) or a diet supplemented with few amino acids. In previous work, a mixed source of protein has been used, mainly from meat (beef, chicken, fish). These types of diets have been criticised because of the potential negative side effects, including our own work on gut health. It might be that alternative vegetable sources of protein could fulfil the diet remit, to be satiating and yet still allow weight loss, and maintain a healthy gut.

Design -within subject, randomised cross-over design after day 3. Each subject acts as their own control and will receive each treatment. 18-20 subjects to participate.

Length of time - Conduct the two nutritional interventions over a period of 14 days, in order to reduce effects due to an acute change in nutritional intake.

PROTOCOL Days 1- 3 - Normal Protein Maintenance diet (NP- MTD, 3 days)

1. st ARM Days 4-17 - randomised to High Protein-Weight loss-Meat (HP-Soya,14 days),
2. nd ARM Days 18-31 - randomised to High Protein-Weight loss-Soya (HP-meat,14 days),

DETAILED DESCRIPTION:
From literature we know that:

* Within-day experiment feeding myco-protein (quorn) versus chicken at lunch resulted in an 18% reduction in evening meal ad libitum intake following the quorn meal (Burley, P. Blundell, 1993, Eur J Clin Nutr, 409-18).
* Feeding casein, soy, pea, wheat gluten, egg albumin, gelatin as part of a mixed meal had no influence on post-lunch satiety (Lang et al.,1998, Am J Clin Nutr., 1197-204).
* Varying protein source (soy, caseine, gelatin) at breakfast meal at 1.8 and 3.6MJ/meal had no impact on 24 hour energy or macronutrient intakes (Lang et al., 1999, Eur J Clin Nutr, 959-65).
* Comparison of mycoprotein and tofu to a chicken preload before lunch indicated that the vegetarian sources were associated with lower food intake at lunch (Williamson et al., 2006, Appetite, 41-8).
* Addition of 25g protein in a liquid format (whey and soy) led to suppression of food intake (pizza meal) 1 hour later, in comparison to water and whey preload.

It is noted that all of these studies, (i) were conducted over a short time period (within day), (ii) none were high-protein weight loss diets (low calorie, high protein), (iii) none compared mixed meat versus vegetable source. It is of interest from both a scientific and public health point of view whether meat and vegetarian sources of protein similarly impact on motivation to eat.

The diets for this study:

* The maintenance diet (MTD) (day 1 - 3) will consist of 15% protein, 30% fat and 55% carbohydrate fed to 1.5 x RMR (resting metabolic rate)
* The high protein (HP) weight loss diet will be fed to 100% resting metabolic rate (RMR) on a 5 day rotation menu, fed as three meals a day, 30% protein, 30% fat and 40% carbohydrate; the meat version will be based on chicken and beef meat; the soya version based on soya protein or soya-tvp (textured vegetable protein).

Soya protein is now widely available as milk (ALPRO), margarine (PURE), enhanced bread (BURGEN), sausages (GRANOSE), bacon (GRANOSE), burgers (GRANOSE), mince (GRANOSE), powered isolate, cheese, cream (SOYA DREAM), yoghurt (ALPRO), chicken-style fillets (GRASSINGTONS).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Overweight or obese (BMI 27+ )
* With no existing medical conditions or medication that could influence appetite or mood.

Exclusion Criteria:

* Diabetes
* Severe gastrointestinal disorders
* Kidney disease
* Thromboembolic or coagulation disease
* Hepatic disease
* Alcohol or any other substance abuse
* Gout
* Eating disorders
* Food allergy
* Unregulated thyroid disease
* Psychiatric disorders (including severe depression, lithium treatment, schizophrenia, severe behavioural disorders)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
appetite control | Every day of the study: From day 1 to 32 inclusive
  * Motivation to eat (VAS) hourly during waking hours up to 6pm in the evening, collected on a hand-help computer
  * Food diary
  * End of day questionnaire on mood

SECONDARY OUTCOMES:
Satiety biomarkers- COMPOSITE MEASURE | test day (day 1, 4, 18, 32 of the study)
  * Subjects will undergo a nutritional challenge on days 4, 18 and 32, where they will attend the Human Nutrition Unit for a meal test (breakfast and lunch, separated by a 5 hr interval) with frequent blood sampling from a cannulae in the arm/hand. Total blood sample collection on each test day will be no more than 120ml per session, collected between 8am and 1pm. Blood samples will be used to measure plasma amino acid concentration, metabolites (e.g. lipids, glucose) and hormones relating to appetite (e.g. PYY). The meal test will consist of their standard meal from their menu.
  * Body composition by bod pod, skinfolds and circumferences
  * Two questionnaires - TFEI (Three-Factor Eating Inventory questionnaire)and DEBQ (Dutch Eating Behaviour) to assess influences on eating
  * Resting metabolic rate using ventilated hood
  * Blood pressure and pulse

OTHER OUTCOMES:
Weight loss | Every day of the study from day 1 to 32 inclusive
  The subjects visited the Human Nutrition Unit at the Rowett Institute of Nutrition and Health (RINH), Aberdeen, United Kingdom daily for the weight measurement, after voiding, while wearing only a previously weighed dressing gown, to the nearest 100 g on a digital scale (DIGI DS-410; CMS Weighing Equipment, London, United Kingdom).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M Johnstone, PhD, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen, Aberdeen, Scotland, UK,; Wendy R Russell, PhD, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen, Aberdeen, Scotland, UK,; Silvia Gratz, PhD, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen, Aberdeen, Scotland, UK,; Graham Horgan, PhD, Principal Investigator — Biomathematics and Statistics Scotland, Aberdeen, Scotland, UK
Locations (1):
- Rowett Institute of Nutrition and Health, University of Aberdeen, Aberdeen, United Kingdom

REFERENCES:
- [Derived] Neacsu M, Fyfe C, Horgan G, Johnstone AM. Appetite control and biomarkers of satiety with vegetarian (soy) and meat-based high-protein diets for weight loss in obese men: a randomized crossover trial. Am J Clin Nutr. 2014 Aug;100(2):548-58. doi: 10.3945/ajcn.113.077503. Epub 2014 Jun 18. PMID 24944057